CLINICAL TRIAL: NCT06638268
Title: Transcatheter AortiC Valve Implantation in AorTic StenosIs CardiogenIc Shock - the TACTICS Study - a Randomized Controlled Trial
Brief Title: Transcatheter AortiC Valve Implantation in AorTic StenosIs CardiogenIc Shock
Acronym: TACTICS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Emil Loldrup Fosbol, Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-24052460
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-09

CONDITIONS: Aortic Stenosis; Cardiogenic Shock
Keywords: Randomized Controlled Trial; Cardiogenic Shock; Aortic Stenosis; Mortality; Frailty; Quality Of Life; Aortic Valve Stenosis; Transcatheter Aortic Valve Replacement; Transcatheter Aortic Valve Implantation
MeSH Terms: conditions — Aortic Valve Stenosis; Shock, Cardiogenic; Frailty

STUDY DESIGN:
Intervention Model Description: Randomized open label trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acute TAVI (Experimental): Acute TAVI within 12 hours.
  Interventions: Procedure: Acute TAVI
- Standard treatment (Active Comparator): TAVI no earlier than 72 hours.
  Interventions: Other: Stabilization and subacute TAVI

INTERVENTIONS:
Procedure: Acute TAVI — TAVI must be performed as soon as possible and within 12 hours of admission to the heart center.
  Arms: Acute TAVI
Other: Stabilization and subacute TAVI — Patients are stabilized according to target parameters. Treatment may include vasopressor, mechanical ventilation, renal replacement therapy, and blood transfusion. TAVI is then performed no earlier than 72 hours of admission to heart center.
  Arms: Standard treatment

SUMMARY:
The goal of this clinical trial is to learn if acute transcatheter aortic valve implantation (TAVI) is superior to standard treatment (stabilization in an intensive care unit and TAVI subsequently) to treat cardiogenic shock in patients with critical severe aortic stenosis.

The main questions it aims to answer are:

• Does acute TAVI increase survival compared with standard treatment?

Participants will:

* Undergo either TAVI within 12 hours after admission or stabilization and TAVI 72 hours or more after admission
* Visit an outpatient clinic and be evaluated for quality of life and heart function

DETAILED DESCRIPTION:
Aortic stenosis (AS) is a condition where the heart's aortic valve narrows. With an estimated prevalence of 12% in individuals aged 75 years and above, it is the most common heart valve disease. The progressive narrowing increases the afterload on the heart, impairing its ability to maintain cardiac output. The end-stage of critical AS is cardiogenic shock (CS) with an incidence of 3.5% to 12%. Without treatment, patients develop acute decompensation, organ failure, and ultimately die.

Guidelines suggest balloon aortic valvuloplasty (BAV), hemodynamic optimization in the intensive care unit and surgical aortic valve replacement or transcatheter aortic valve implantation (TAVI) when the patient is stable. Even with BAV, the 30-day mortality is 33%-47% and a 1-year mortality is 70%. Further, the BAV procedure is associated with only a minor and likely temporary reduction in afterload due to elastic valvular tissue. Furthermore, the BAV procedure has been abandoned as a routine intervention in these patients due to a series of patients having limited immediate clinical response, a risk of deterioration and no impact on overall mortality risk. Moreover, most patients with critical AS in CS are not candidates for surgical aortic valve replacement because of increased peri-operative risk of morbidity and mortality.

Despite the recommendation on TAVI under stable conditions, an acute TAVI may be efficient in afterload reduction and more efficient than the limited and transient effects of BAV. TAVI has become an attractive alternative to surgery and BAV because of the less invasive nature of this procedure, yet permanent result (compared with BAV). It is already approved for the treatment of AS irrespective of CS status. This raises the question:

"Should acute TAVI be the new preferred treatment strategy in AS patients in Cardiogenic shock?"

In this randomized controlled trial, we will include patients with severe aortic stenosis and cardiogenic shock. Patients will undergo either acute TAVI or standard treatment (stabilization in a cardiac intensive care unit and subsequently TAVI) in a 1:1 ratio. Outcomes are evaluated 90 days after randomization and comprise days alive out of hospital, mortality, cardiac function, renal function, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Aortic valve area less than 1cm2

AND

Cardiogenic Shock defined as:

* Peripheral signs of tissue hypoperfusion (arterial blood lactate ≥2.5mmol/l) AND
* Systolic blood pressure < 100 mmHg and/or need for vasopressor therapy (dopamine/ norepinephrine or epinephrine) AND
* Left ventricular ejection fraction ≤ 45%

OR

- Syncope/resuscitation (mechanical ventilation)

Exclusion Criteria:

* Intracranial hemorrhage < 1 month ago
* Remaining life-expectancy < 6 month due to other cause
* Body mass index <15 OR > 40
* Clinical frailty score ≥6 before present worsening
* Severe lung disease (forced expiratory volume in 1 second OR diffusion capacity of the lungs for carbon monoxide < 25 of expected)
* Unsuitable for TAVI prior to screening

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-25 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Days alive out of hospital | 90 days post-randomization
  Days alive out of hospital

SECONDARY OUTCOMES:
Mortality | 90 days post-randomization
  Rate of all-cause mortality
LVEF | 90 days post-randomization
  Left ventricular ejection fraction assessed with transthoracic echocardiography
Clinical Frailty Scale | 90 days post-randomization
  The Clinical Frailty Scale (CFS) is a tool used to assess a patient's level of frailty. The CFS ranges from 1 to 9, with higher scores indicating greater frailty.
EQ-5D-5L | 90 days post-randomization
  The EQ-5D-5L is a standardized instrument used to measure health-related quality of life. It is designed for use in clinical settings, research, and health evaluations, and provides a simple, yet comprehensive measure of a patient's overall health status. The "5D" refers to the five dimensions of health that it assesses, and the "5L" refers to the five levels of severity within each dimension.
N-terminal-pro-brain- natriuretic peptide levels | 90 days post-randomization
  Meassured in a blood sample
eGFR | 90 days post-randomization.
  Estimated glomerular filtration rate in mL/min/1.73m2 meassured in a blood sample.

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Rigshospitalet Copenhagen University Hospital, Copenhagen O
  - Odense University Hospital, Odense C

IPD SHARING:
Plan to Share IPD: No